CLINICAL TRIAL: NCT04209868
Title: Preoperative Paravertebral Block in Cancer Surgery of the Lung: ParaSOL a Prospective Randomized Controlled Clinical Trial
Brief Title: Preoperative Paravertebral Block in Cancer Surgery of the Lung
Acronym: ParaSOL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 244680
Record Dates: First submitted 2019-11-21; First posted 2019-12-24 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Thoracic Neoplasm; Chronic Pain Post-Procedural; Acute Post-thoracotomy Pain; Anesthesia, Local
MeSH Terms: conditions — Thoracic Neoplasms | interventions — Injections; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study will be conducted at Guy's Hospital, London, United Kingdom (UK), a large tertiary thoracic centre for London, Sussex, Kent and Berkshire. In 2015, 459 lung cancer resection operations were performed; 8% of all lung cancer resections in England.
  Criteria for discontinuation/withdrawal or modifying allocated treatment:
  * Participant request to withdraw from the study.
  * Intraoperative identification of infection/tumour in paravertebral space
  Patient recruitment Eligible patients will be identified in the catchment outpatient clinics 4-6 weeks before surgery. The participant information sheet (PIS) will be introduced in the standard surgical booklet given by the surgeon. At the preoperative assessment clinic 2-3 weeks before surgery, a face-to-face discussion with the research nurse will support the PIS; the opportunity to ask any questions and contact a PPI (Patient and Public Involvement) representative and will be given. Written informed consent will be obtained.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomised on the day of surgery to the 'pre-PVB LA' or 'pre-PVB saline' arm, by a study investigator, with a 1:1 randomisation ratio using 'Sealed Envelope' (www.sealedenvelope.com) online software. Each subject will receive a unique randomization code in an envelope that will only be opened during the preparation of the pre-PVB injectate.
  A non-blinded research nurse, will prepare the pre-PVB injectate in a standard syringe according to the allocation, labelled by participant number, in a theatre location concealed from the operating room and staff.
  The anaesthetist, the surgeon and theatre team, recovery staff, and the researchers performing all the outcome assessments will be separate and blinded to the group allocation. The PVB catheter will be taped as normal before connecting the post-PVB LA infusion pump.
  We have elected to perform an interventional placebo intervention as opposed to a sham control to minimize observer bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-PVB with saline (Placebo Comparator): Placebo (20ml Saline) pre-PVB performed post-induction and pre-incision.
  Interventions: Drug: 0.9% Sodium Chloride 20mL Injection
- Pre-PVB with 0.5% Levo-bupivacaine (Experimental): 20ml 0.5% Levo-bupivacaine pre-PVB performed post-induction and pre-incision.
  Interventions: Drug: Levo-Bupivacaine Hydrochloride (HCl) 0.5 % in 20mL Injection

INTERVENTIONS:
Drug: Levo-Bupivacaine Hydrochloride (HCl) 0.5 % in 20mL Injection — As per arm description
  Arms: Pre-PVB with 0.5% Levo-bupivacaine
Drug: 0.9% Sodium Chloride 20mL Injection — As per arm description
  Arms: Pre-PVB with saline

SUMMARY:
The investigators aim to determine whether ultrasound-guided preemptive paravertebral blockade (PVB) local anaesthetic (pre-PVB LA), administered in addition to the post-operative PVB (post-PVB) local anaesthetic (LA) infusion, reduces acute postoperative pain, opioid requirement, chronic pain, and improves surgical recovery, in thoracoscopic surgery for lung cancer.

DETAILED DESCRIPTION:
In the UK, there has been an increase in lung cancer operations, especially in high risk and elderly patients, improving survival from 10.6% in 2008 to 15.1% in 2013. Lung cancer surgery is associated with severe acute pain, a high incidence of respiratory complications and chronic post-surgical pain. Severe acute postoperative pain is a strong predictor of CPSP. The improvement of perioperative outcomes in elderly patients, the benefits of regional anaesthesia and reduction of chronic pain are investigative priorities of the Anaesthesia and Perioperative Care Setting Partnership.

Enhanced recovery strategies include video-assisted thoracoscopic surgery (VATS), a minimally invasive alternative to open thoracotomy, which may be associated with less postoperative pain. Regional anaesthesia, by thoracic epidural analgesia (TEA) or PVB, is superior to systemic opioids in reducing acute pain after thoracotomy surgery.

Preemptive analgesia describes the aim of minimizing central spinal pain transmission by noxious stimuli arising from events at surgery, by administering an analgesic technique prior to surgical incision. Regional blockade affects central sensitization, allowing analgesia to outlast the pharmacological sensory blockade.

Compared to TEA initiated after surgery, acute pain severity is reduced by preemptive TEA. There are conflicting reports on the benefit of preemptive analgesia in other types of surgery, but TEA and PVB may prevent CPSP in thoracotomy and breast surgery. Some small studies have shown that pre-PVB reduces acute postoperative pain.

Paravertebral blockade is known to be as effective as TEA for acute postoperative analgesia following thoracic surgery, whilst having a lower incidence of pulmonary complications, hypotension and nausea. It is conventional practice in many centres for the surgical administration and placement of a catheter at the end of surgery for postoperative LA infusion (post-PVB) as the sole method of regional analgesia. Preoperative PVB is less common: anaesthetists may use a landmark technique, single or multiple injections and different volumes/strengths of LA.

Ultrasound guidance for pre-PVB injection increases accuracy. In an audit using this technique with post-PVB compared to post-PVB only, the investigators demonstrated reduced pain numerical rating scale (NRS) scores in elective VATS patients, (mean NRS at 24h 2.5 vs 4.5), and a reduction in the proportion of patients who experienced moderate-to-severe pain of NRS≥ 3 from 83% to 50% at 24h.

The investigators therefore aim to evaluate the contribution of ultrasound-guided pre-PVB, administered in addition to the post-PVB LA infusion, in reducing the severity of acute postoperative pain, perioperative opioid requirement, development of CPSP, and improving patient outcome in lung cancer patients undergoing VATS.

ELIGIBILITY:
Inclusion Criteria:

* Elective radical primary lung cancer VATS surgery for single lobectomy
* American Society of Anesthesiology (ASA) I-III
* Age ≥18

Exclusion Criteria:

* Planned open thoracotomy, wedge resection, bilobectomy, pneumonectomy, chest wall resection or total pleurectomy
* Local anaesthetic or opioid allergy
* Coagulation disorders
* Inability to comply with study questionnaire completion
* Pre-existing pain in chest area or pre-existing pain conditions
* Local infection/tumour at proposed PVB site
* Previous lung surgery
* Planned surgery within 3 months of the primary lung resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Moderate-to-severe pain Numerical Rating Scale (NRS) >/=3 | 1 day
  The proportion of patients with clinical relevant moderate-to-severe pain (NRS>/=3) related to the surgical site at rest at 24 hours.

SECONDARY OUTCOMES:
Acute postoperative pain related to the surgical site as measured by a numerical rating scale (NRS) at rest and on coughing. | 1 hour
  Acute postoperative pain related to the surgical site as measured by a numerical rating scale (NRS) at rest and on coughing, preoperatively, and after arrival in recovery at 1, 6, 24 and 48 hours
Acute postoperative pain related to the surgical site as measured by a numerical rating scale (NRS) at rest and on coughing. | 6 hours
  Acute postoperative pain related to the surgical site as measured by a numerical rating scale (NRS) at rest and on coughing, preoperatively, and after arrival in recovery at 1, 6, 24 and 48 hours
Acute postoperative pain related to the surgical site as measured by a numerical rating scale (NRS) at rest and on coughing. | 24 hours
  Acute postoperative pain related to the surgical site as measured by a numerical rating scale (NRS) at rest and on coughing, preoperatively, and after arrival in recovery at 1, 6, 24 and 48 hours
Acute postoperative pain related to the surgical site as measured by a numerical rating scale (NRS) at rest and on coughing. | 48 hours
  Acute postoperative pain related to the surgical site as measured by a numerical rating scale (NRS) at rest and on coughing, preoperatively, and after arrival in recovery at 1, 6, 24 and 48 hours
Cumulative morphine requirement | 48 hours
  Cumulative morphine requirement over 48 hours post arrival in recovery
Time to first mobilization | 3 days
  Time to first mobilization (walking 50 metres without the aid of another person), measured at baseline pre-operatively and postoperatively on daily assessment.
Incidence of in-hospital complications | 3 days
  Incidence of in-hospital complications (Atrial Fibrillation (AF), Myocardial Infarction (MI), unplanned ICU admission) and respiratory complications, as defined by the Melbourne Group Scale.
Length of hospital stay | 3 days
  Length of hospital stay (in days)
Quality of Life (QoL) score | Pre-operative and at 3 and 6 months post-operatively
  Quality of Life (QoL) score as measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) version 3
Presence of chronic post-surgical pain | Measured at 3 and 6 months post-operatively
  Presence of chronic post-surgical pain (CPSP) (binary yes/no) fulfilling CPSP criteria
Presence of chronic post-surgical pain | Measured at 3 and 6 months post-operatively
  Presence of chronic post-surgical pain assessed by the Brief Pain Inventory Short Form (BPI-SF)
Presence of chronic post-surgical pain | Measured at 3 and 6 months post-operatively
  Presence of chronic post-surgical pain assessed by as defined by the Melbourne Group Scale

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Ong, Study Chair — Guys & St Thmas' NHS Foundation Trust
Locations (1):
- Guy's Hospital, Great Maze Pond, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT04209868/Prot_SAP_001.pdf